CLINICAL TRIAL: NCT06611618
Title: Analisi Della Perdita di Forza e Potenza Muscolare e Del Degrado Del Controllo Motorio Per la Predizione Delle Cadute in Una Popolazione Affetta da Artrosi di Ginocchio
Brief Title: Analysis of the Loss of Muscle Force, Muscle Power and Motor Control Degradation to Predict the Risk of Falls in Patients With Knee Osteoarthritis
Acronym: PowerAGING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE-AVEC 204/2024/Sper/IOR
Record Dates: First submitted 2024-09-17; First posted 2024-09-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis (Knee OA); Falls Prevention
Keywords: Falls prevention; Knee osteoarthritis; Muscle power; Muscle force; Motor control degradation; digital twins; IMU; mobility monitoring; MRI
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee Osteoarthritis (Experimental): Elderly patients with knee osteoarthritis, without a history of falls (in the 12 months prior to enrollment).
  All subjects will be followed up for 24 months, every 6 months. Muscle force and power assessments, plus a home-based mobility monitoring, will be performed at all visits. Full lower limb MRI and a gait assessment will be performed at first and last visit.
  Interventions: Other: Muscle power assessment; Other: Muscle force assessment; Other: Home-based mobility monitoring; Diagnostic Test: Magnetic Resonance Imaging; Other: Gait assessment

INTERVENTIONS:
Other: Muscle power assessment — Isokinetic dynamometry test Stair ascent/descent on instrumented stairs
Other: Muscle force assessment — Isometric dynamometry (Maximal Voluntary Isometric Contraction)
Other: Home-based mobility monitoring — Mobility monitoring with wearable sensors
Diagnostic Test: Magnetic Resonance Imaging — Full lower limb MRI
Other: Gait assessment — Motion capture, surface EMG and gorund reaction force data

SUMMARY:
The twofold goal of this study is to understand the link between muscle power, muscle strength, and muscle control degradation with the risk of falling, and to develop a framework for the comprehensive and quantitative assessment of muscle power (and strength) in an elderly population of patients with knee osteoarthritis, who are at higher risk of falling. The main question it aims to answer is:

● Are muscle power and motor control degradation better predictors of falls than muscle strength in the aging population?

Participants will undergo:

* Muscle force assessment on a dynamometer
* Muscle power assessment on a dynamometer and on isntrumented stairs
* Home-based mobility monitoring
* Full lower limb MRI acquisition
* Gait assessment

DETAILED DESCRIPTION:
Falls are a critical yet common event among the elderly, with huge societal and economic impact (reduced quality of life and high costs for the healthcare system). Experimental measures to quantify the residual muscle strength and power may provide useful information to predict the risk of falls in the elderly. Isometric and isokinetic muscle contractions, performed on a dynamometer or during functional tasks can be collected, together with electromyography (to assess muscle activity) and imaging data (to quantify and characterize muscular tissue).

Such data can be collected at different time points to monitor subjects over time, and to inform virtual representation of the human musculoskeletal system (digital twins) to identify possible motor control deficits. Moreover, this same information can be used to better characterize/assess elder individuals at risk of falling (e.g., subjects with knee osteoarthritis), to prevent future falls.

All subjects enrolled in the PowerAGING study will be followed up for 24 months (5 visits in total: M0, M6, M12, M18 and M24 follow-up). At each visit, a series of experimental tests to quantify muscle power and muscle force, as well as a home-based mobility assessment (via single inertial sensor worn for 5 consecutive days), will be performed. In addition, only at start and end, the subjects will undergo a full lower limb MRI and a gait assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 80 years
* Kellgren score II e III
* No history of falls in the last 12 months

Exclusion Criteria:

* Any musculoskeletal, neurological, rheumatic or tumoral diseases
* Dementia
* Diabetes
* Inguinal or abdominal hernia
* Severe Hypertension (Level 3)
* Severe Cardio-pulmonary insufficiency
* Diagnosis of Osteonecrosis in the lower limb joints
* Pathologies or physical conditions incompatible with the use of magnetic resonance imaging and electrostimulation (i.e., active and passive implanted biomedical devices, epilepsy, severe venous insufficiency in the lower limbs)
* Previous interventions or traumas to the joints of the lower limb

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Muscle volumes | From baseline (Day 0) to last visit (Month 24)
Maximal muscle force | At baseline (Day 0) and all follow-up visits (Month 6, Month 12, Month 18, Month 24)
  Maximal Isometric muscle force from dynamometry test
Muscle power | At baseline (Day 0) and all follow-up visits (Month 6, Month 12, Month 18, Month 24)
  Assessed on the dynamometer and during dynamic tasks
Muscle activations | At baseline (Day 0) and all follow-up visits (Month 6, Month 12, Month 18, Month 24)
  From surface EMG data collected on the dynamometer and during dynamic tasks (gait assessment and stair ascent/descent)
Digital Mobility Outcomes | At baseline (Day 0) and all follow-up visits (Month 6, Month 12, Month 18, Month 24)
  Qualitative and quantiative measures of real-world mobility (e.g., gait speed, stride length)
Musculoskeletal model predictions | At baseline (Day 0) and all follow-up visits (Month 6, Month 12, Month 18, Month 24)
  Estimates of muscle force and knee joint contact forces

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy